CLINICAL TRIAL: NCT00598754
Title: Diagnostic Two and Three Dimensional Echocardiography Study Protocol
Brief Title: Diagnostic Three Dimensional Echocardiography Study Protocol
Status: Withdrawn | Type: Observational
Why Stopped: Funding issues
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Space Biomedical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NSBRI NCC9-59-172 #1; IRB 4401; Cardiac mass regression; 3 dimensional echocardiography; Project # SMS004-004
Record Dates: First submitted 2007-12-20; First posted 2008-01-22 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: Aortic valve stenosis; Aortic valve insufficiency; Two dimensional echocardiography; Three dimensional echocardiography
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to perform ground-based research to study what happens to the heart muscle in space. People who have problems with their aortic valve have an increase in the amount of muscle in the left ventricle of the heart. After valve surgery, the amount of muscle should decrease and return to normal. Astronauts lose heart muscle mass during space flight. Our study will look at these changes in your heart, which we believe are similar to what happens during long term space travel.

This study will look at the accuracy of three dimensional ultrasound imaging (echo) in monitoring the changes in heart size and function following aortic valve replacement. We are studying ways to prevent health-related problems that men and women will face on long-duration space missions.

The hypothesis is that serial two dimensional and three dimensional echo will show accurate changes in the left ventricle mass and volume following aortic valve replacement for aortic stenosis or regurgitation

DETAILED DESCRIPTION:
Diagnostic Three Dimensional Echocardiography Study Protocol

A. Aims The overall purpose of this study is to perform ground-based research, development, and validation aimed at optimizing diagnostic ultrasound in manned spaceflight, with the following unifying hypothesis: Serial 3D ultrasound examinations will enhance diagnostic capabilities in manned spaceflight.

Specific Aims:

1. To optimize acquisition methods for 3D sonography using reconstruction and real-time techniques
2. To determine the utility of serial 3D ultrasound examinations in identifying renal calculi and their complications including the development and resolution of hydronephrosis and calyceal dilatation.
3. To determine the utility of serial 2D and 3D ultrasound examinations in demonstrating cardiac remodeling (changes in cardiac dimensions, volume, mass and function) and defining its determinants after left ventricular unloading following aortic valve replacement for aortic stenosis or regurgitation.
4. To determine whether changes in plasma BNP levels accurately reflect changes in LV mass and volume.

Hypotheses:

1. Serial 3D ultrasound examinations will allow accurate diagnosis of nephrolithiasis and tracking of complications including hydronephrosis and calyceal dilatation
2. Serial 2D and 3D ultrasound will allow accurate tracking of changes in LV mass and volume following aortic valve replacement (AVR) for aortic stenosis or regurgitation.
3. Changes in plasma BNP levels will fall in proportion to the decrease in LV mass and volume.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgery for aortic stenosis or aortic regurgitation

Exclusion Criteria:

* Previous open heart surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming to Cleveland Clinic to have surgery for aortic stenosis or aortic insufficiency.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2001-06; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic 2D and 3D echocardiography | 6 - 12 months

SECONDARY OUTCOMES:
BNP levels | 6-12 months
MRI | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jim D Thomas, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No